CLINICAL TRIAL: NCT05162417
Title: Efficacy of Some Different Photosensitizers in Photodynamic Inactivation of Periodontal Pathogens:A Randomized Clinical Trial
Brief Title: Photodynamic in Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Sarhang Gul, Asst. Prof., University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55/21
Record Dates: First submitted 2021-11-29; First posted 2021-12-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Diseases; Periodontal Pocket
Keywords: Probing Pocket depth; phhotosensitizers
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket | interventions — Methylene Blue; Tolonium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): patient in this arm will receive scaling and root planning treatment only.
- Test group (toluidine Blue O) (Experimental): patients in this arm will receive Toluidine Blue O as an adjunctive to scaling and root planing.
  Interventions: Other: Toluidine Blue O
- Methylene blue (Experimental): Patients will receive Methylene blue as adjunctive to scaling and root planning.
  Interventions: Other: Methylene Blue

INTERVENTIONS:
Other: Methylene Blue — 1mg/ml of Methylene as a solution will be used two times, first immediately after scaling and root planning, second after two weeks of the first treatment.
  Arms: Methylene blue
Other: Toluidine Blue O — 1mg/ml of Toluidine blue o as a solution will be used two times, first immediately after scaling and root planning, second after two weeks of the first treatment.
  Arms: Test group (toluidine Blue O)

SUMMARY:
Dental biofilm is a primary etiological factor for periodontal diseases.(1) The bacterial biofilm would induce recruitment of leucocytes, neutrophils, and T lymphocytes and the secretion of antibodies, lipopolysaccharides, and chemical inflammatory mediators such as cytokines and chemokines.(2) Thus, periodontal diseases can cause tissue destruction and results in deterioration of clinical parameters measures such as periodontal pockets depth, clinical attachment loss, bleeding on probing, bone destruction, and resulting ultimately in tooth loss.(3)

DETAILED DESCRIPTION:
Mechanical scaling and polishing are the conventional methods in treating periodontal diseases; however, due to difficulties in access to the irregular and furcation areas, it is impossible to be used as a sole means for calculus and bacterial deposit removal.(4) For this reason, adjunctive aids like systemic and local antibiotics are necessary to be administrated However, they have many adverse effects.(5) Another adjunctive aid like antibacterial photodynamic therapy (APDT), has been introduced to periodontology to achieve bacterial eradication, with minimum side effects.(6) APDT involves using visible light with an appropriate wavelength to kill microorganisms with a photosensitizing drug.(7) APDT could be an adjunctive aid to mechanical debridement in eliminating key periodontal pathogens. This therapy was specified as an oxygen-dependent photochemical reaction upon light-mediated activation of photosensitizing materials leading to cytotoxic reactive oxygen species (ROS) generation, predominantly singlet oxygen.(8) The activity of APDT is dependent on the combination of a non-toxic photosensitizer and a specific wavelength of visible light, which is activated and can promote a phototoxic response in the presence of ambient oxygen.(9) APDT is characterized by ROS generation by PSs in response to photo illumination, which later causes cell death.(6)

ELIGIBILITY:
Inclusion Criteria:

* Each patient should have at least four teeth with a probing depth ≥of 5mm.
* Patients with good domestic oral hygiene will be include (documented with a full mouth plaque index of ≤ 30% before starting the clinical trial)

Exclusion criteria:

* Patients receiving periodontal therapy and/or antibiotics within the previous six months
* Patients with diseases or medication with an inhibitory or promoting effect on periodontal healing, including anticoagulants, anti-inflammatories.
* Pregnant or nursing women
* Patients allergic to the test product will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in probing pocket depth | At the base line and three months
  millimetre
Change in clinical attachment loss | At the base line and three months
  millimeter

SECONDARY OUTCOMES:
Change in bleeding on Probing | at base line and 3 month
  present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Sarhang S. Gul, PhD, Principal Investigator — College of Dentistry, University of Sulaimani
Locations (1):
- College of Dentistry, University of Sulaimani, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request following publication by principal investigators
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: The data will be available upon reasonable request.
URL: https://sites.google.com/a/univsul.edu.iq/school-of-dentistry/

REFERENCES:
- [Background] Larsen T, Fiehn NE. Dental biofilm infections - an update. APMIS. 2017 Apr;125(4):376-384. doi: 10.1111/apm.12688. PMID 28407420
- [Background] Cekici A, Kantarci A, Hasturk H, Van Dyke TE. Inflammatory and immune pathways in the pathogenesis of periodontal disease. Periodontol 2000. 2014 Feb;64(1):57-80. doi: 10.1111/prd.12002. PMID 24320956
- [Background] Kinane DF, Stathopoulou PG, Papapanou PN. Periodontal diseases. Nat Rev Dis Primers. 2017 Jun 22;3:17038. doi: 10.1038/nrdp.2017.38. PMID 28805207
- [Background] Shrivastava D, Natoli V, Srivastava KC, Alzoubi IA, Nagy AI, Hamza MO, Al-Johani K, Alam MK, Khurshid Z. Novel Approach to Dental Biofilm Management through Guided Biofilm Therapy (GBT): A Review. Microorganisms. 2021 Sep 16;9(9):1966. doi: 10.3390/microorganisms9091966. PMID 34576863
- [Background] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- [Background] Carrera ET, Dias HB, Corbi SCT, Marcantonio RAC, Bernardi ACA, Bagnato VS, Hamblin MR, Rastelli ANS. The application of antimicrobial photodynamic therapy (aPDT) in dentistry: a critical review. Laser Phys. 2016 Dec;26(12):123001. doi: 10.1088/1054-660X/26/12/123001. Epub 2016 Nov 9. PMID 29151775
- [Background] Kharkwal GB, Sharma SK, Huang YY, Dai T, Hamblin MR. Photodynamic therapy for infections: clinical applications. Lasers Surg Med. 2011 Sep;43(7):755-67. doi: 10.1002/lsm.21080. PMID 22057503
- [Background] Kashef N, Huang YY, Hamblin MR. Advances in antimicrobial photodynamic inactivation at the nanoscale. Nanophotonics. 2017 Aug;6(5):853-879. doi: 10.1515/nanoph-2016-0189. Epub 2017 Aug 1. PMID 29226063
- [Background] Liu Y, Qin R, Zaat SAJ, Breukink E, Heger M. Antibacterial photodynamic therapy: overview of a promising approach to fight antibiotic-resistant bacterial infections. J Clin Transl Res. 2015 Dec 1;1(3):140-167. eCollection 2015 Dec 30. PMID 30873451
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/28407420/
- See also: pubmed resource — http://pubmed.ncbi.nlm.nih.gov/24320956/
- See also: pubmed resource — http://pubmed.ncbi.nlm.nih.gov/28805207/
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/34576863/
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/33197289/
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/29151775/
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/22057503/
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/29226063/
- See also: pubmed resource — https://pubmed.ncbi.nlm.nih.gov/30873451/